CLINICAL TRIAL: NCT02966535
Title: The Effect of Prolonged Inspiratory Time on Gas Exchange During Robot-assisted Laparoscopic Surgery With Steep Trendelenburg Position : A Crossover Randomized Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Won Ho Kim, MD, Clinical Associate Professor, Seoul National University Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 1609-102-793
Record Dates: First submitted 2016-11-13; First posted 2016-11-17 (Estimated); Last update posted 2019-03-14 (Actual); Status verified 2017-09

CONDITIONS: Prostatic Neoplasm; Urinary Bladder Neoplasm
MeSH Terms: conditions — Prostatic Neoplasms; Urinary Bladder Neoplasms

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1:2, 1:1 group (Experimental): Inspiratory to expiratory time ratio (I:E ratio) of 1:2 during the first one hour of laparoscopy and then switched to I:E ratio of 1:1 during the rest time of laparoscopy.
  Interventions: Device: Adjustment of Mechanical Ventilator Inspiratory to expiratory time ratio (1:2 to 1:1)
- 1:1, 1:2 group (Active Comparator): Inspiratory to expiratory time ratio (I:E ratio) of 1:1 during the first one hour of laparoscopy and then switched to I:E ratio of 1:2 during the rest time of laparoscopy.
  Interventions: Device: Adjustment of Mechanical Ventilator Inspiratory to expiratory time ratio (1:1 to 1:2)

INTERVENTIONS:
Device: Adjustment of Mechanical Ventilator Inspiratory to expiratory time ratio (1:2 to 1:1) — Adjustment of Mechanical Ventilator Inspiratory to expiratory time ratio (1:2 to 1:1)
  Arms: 1:2, 1:1 group
Device: Adjustment of Mechanical Ventilator Inspiratory to expiratory time ratio (1:1 to 1:2) — Adjustment of Mechanical Ventilator Inspiratory to expiratory time ratio (1:1 to 1:2)
  Arms: 1:1, 1:2 group

SUMMARY:
Gas exchange disturbance frequently occurs in steep Trendelenburg position during robot-assisted laparoscopic prostatectomy or cystectomy. Due to increased intrathoracic pressure and absorbed carbon dioxide (CO2) gas insufflated into abdominal cavity, hypercapnia as well as hypoxia may occur. Inverse ratio ventilation or prolonged inspiratory time during mechanical ventilation has been reported to be improve gas exchange in adult respiratory distress syndrome. The investigators attempt to test the hypothesis that prolonged inspiratory time may improve the gas exchange during robot-assisted laparoscopic urologic surgery.

DETAILED DESCRIPTION:
Gas exchange disturbance frequently occurs in steep Trendelenburg position during robot-assisted laparoscopic prostatectomy or cystectomy. Due to increased intrathoracic pressure and absorbed CO2 gas insufflated into abdominal cavity, hypercapnia as well as hypoxia may occur. Inverse ratio ventilation or prolonged inspiratory time during mechanical ventilation has been reported to be improve gas exchange in adult respiratory distress syndrome. The investigators attempt to test the hypothesis that prolonged inspiratory time (I:E ratio = 1:1) may improve the gas exchange during robot-assisted laparoscopic urologic surgery.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists physical status class I-II and scheduled for an elective robot-assisted laparoscopic radical prostatectomy or robot-assisted laparoscopic radical cystectomy
* Patients who voluntarily decides to participate in the trial and has agreed in written informed consent

Exclusion Criteria:

* Patients with the anatomical abnormalities of respiratory system(abnormal airway anatomy, severe scoliosis, post-pneumonectomy state), severe chronic respiratory diseases, chronic obstructive pulmonary disease (COPD), asthma, heart failure, obesity ( Body Mass Index [BMI] > 30kg/m2), severe hepatic failure or renal failure

Ages: 20 Years to 90 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
PaCO2 (mmHg) in the patient's arterial blood gas analysis | 60 min after the initiation of pneumoperitoneum with steep Trendelenburg positioning
  PaCO2 (arterial partial pressure of carbon dioxide)

SECONDARY OUTCOMES:
PaCO2 (mmHg) in the patient's arterial blood gas analysis | 5 minutes after anesthesia induction
  PaCO2 (arterial partial pressure of carbon dioxide)
PaO2 (mmHg) in the patient's arterial blood gas analysis | 5 minutes after anesthesia induction
  PaO2 (arterial partial pressure of oxygen)
PaO2 (mmHg) in the patient's arterial blood gas analysis | 60 minutes after anesthesia induction
  PaO2 (arterial partial pressure of oxygen)
PaCO2 (mmHg) in the patient's arterial blood gas analysis | 120 minutes after anesthesia induction
  PaCO2 (arterial partial pressure of carbon dioxide)
PaO2 (mmHg) in the patient's arterial blood gas analysis | 120 min after the initiation of pneumoperitoneum with steep Trendelenburg positioning
  PaO2 (arterial partial pressure of oxygen)
PaCO2 (mmHg) in the patient's arterial blood gas analysis | 10 min after restoration of supine position
  PaCO2 (arterial partial pressure of carbon dioxide)
PaO2 (mmHg) in the patient's arterial blood gas analysis | 10 min after restoration of supine position
  PaO2 (arterial partial pressure of oxygen)
Respiratory compliance (Static, Dynamic) | 5 minutes after anesthesia induction
  Static compliance = exhaled tidal volume / (plateau pressure - PEEP), Dynamic compliance = Exhaled tidal volume / (PIP - PEEP)
Respiratory compliance (Static, Dynamic) | 60 min after the initiation of pneumoperitoneum with steep Trendelenburg positioning
  Static compliance = exhaled tidal volume / (plateau pressure - PEEP), Dynamic compliance = Exhaled tidal volume / (PIP - PEEP)
Respiratory compliance (Static, Dynamic) | 120 min after the initiation of pneumoperitoneum with steep Trendelenburg positioning
  Static compliance = exhaled tidal volume / (plateau pressure - PEEP), Dynamic compliance = Exhaled tidal volume / (PIP - PEEP)
oxygen index | 5 minutes after anesthesia induction
  oxygen index calculated by PaO2/inspired oxygen fraction
oxygen index | 60 min after the initiation of pneumoperitoneum with steep Trendelenburg positioning
  oxygen index calculated by PaO2/inspired oxygen fraction
oxygen index | 120 min after the initiation of pneumoperitoneum with steep Trendelenburg positioning
  oxygen index calculated by PaO2/inspired oxygen fraction
Alveolar-arterial oxygen difference | 5 minutes after anesthesia induction
Alveolar-arterial oxygen difference | 60 min after the initiation of pneumoperitoneum with steep Trendelenburg positioning
Alveolar-arterial oxygen difference | 120 min after the initiation of pneumoperitoneum with steep Trendelenburg positioning

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] De Carlo F, Celestino F, Verri C, Masedu F, Liberati E, Di Stasi SM. Retropubic, laparoscopic, and robot-assisted radical prostatectomy: surgical, oncological, and functional outcomes: a systematic review. Urol Int. 2014;93(4):373-83. doi: 10.1159/000366008. Epub 2014 Sep 23. PMID 25277444
- [Background] Gainsburg DM. Anesthetic concerns for robotic-assisted laparoscopic radical prostatectomy. Minerva Anestesiol. 2012 May;78(5):596-604. Epub 2012 Mar 13. PMID 22415437
- [Background] Kim MS, Kim NY, Lee KY, Choi YD, Hong JH, Bai SJ. The impact of two different inspiratory to expiratory ratios (1:1 and 1:2) on respiratory mechanics and oxygenation during volume-controlled ventilation in robot-assisted laparoscopic radical prostatectomy: a randomized controlled trial. Can J Anaesth. 2015 Sep;62(9):979-87. doi: 10.1007/s12630-015-0383-2. Epub 2015 Apr 14. PMID 25869025